CLINICAL TRIAL: NCT04594824
Title: Defining Reference Ranges for Cerebral Oxygenation In Neonates (COIN) During Immediate Neonatal Transition After Birth - a Prospective Observational Study
Brief Title: Defining Reference Ranges for Cerebral Oxygenation In Neonates (COIN) During Immediate Neonatal Transition After Birth
Acronym: COIN
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 32-320 ex 19/2
Record Dates: First submitted 2020-10-16; First posted 2020-10-20 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Neonatal Adaptation
Keywords: percentile; cerebral oxygenation; neonate; immediate after birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Term neonates
  Interventions: Other: No Intervention
- Preterm neonates
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — no intervention

SUMMARY:
Especially in neonates non-invasive methods are required for monitoring the complex changes during immediate transition after birth to improve assessment of neonate and eventually resuscitation. During this period especially, the brain is vulnerable and monitoring the brain and possible influencing factors of cerebral oxygenation and perfusion are of great interest. To initiate and guide therapies based on cerebral oxygenation, it is important to define reference ranges.

ELIGIBILITY:
Inclusion Criteria:

* Term and preterm neonates observed routinely at the resuscitation desk
* Decision to conduct full life support
* Written informed consent
* Neonates who require no respiratory or medical support

Exclusion Criteria:

* No decision to conduct full life Support
* No written informed consent
* Congenital malformation
* Neonates who require respiratory and/ or medical support

Ages: 0 Minutes to 15 Minutes | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Neonates immediatley after birth
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
Change of cerebral tissue oxygen saturation (crSO2) level | At each minute from minute 1 to minute 15 after birth
  To measure cerebral oxygenation with Root (O3 regional oxymetry, Masimo, USA) non-invasively and continuously during the first 15 minutes after birth and establish the reference ranges in term and preterm neonates.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Neonatology, Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Undecided